CLINICAL TRIAL: NCT02103478
Title: A Phase1-2 Pharmacokinetic Guided Dose-Escalation and Dose-Confirmation Study of ASTX727, a Combination of the Oral Cytidine Deaminase Inhibitor (CDAi) E7727 With Oral Decitabine in Subjects With Myelodysplastic Syndromes (MDS)
Brief Title: Pharmacokinetic Guided Dose Escalation and Dose Confirmation With Oral Decitabine and Oral Cytidine Deaminase Inhibitor (CDAi) in Patients With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-01
Record Dates: First submitted 2014-03-20; First posted 2014-04-04 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndrome; MDS
Keywords: Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — cedazuridine; Decitabine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 Dose Escalation (Experimental): Starting cohort was administered 40 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  Interventions: Drug: ASTX727 Dose Escalation
- Phase 2 Dose Confirmation (Experimental): Participants were randomized in a 1:1 ratio to receive either oral cedazuridine (E7727) (100 mg) + decitabine (35 mg) capsules Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) or the converse. In Courses ≥ 3, participants received cedazuridine and decitabine capsules Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
  Interventions: Drug: ASTX727 Dose Confirmation
- Phase 2 Fixed-Dose Combination (Experimental): Participants were randomized in a 1:1 ratio to receive either the fixed-dose combination (FDC) tablet (100 mg cedazuridine (E7727)/35 mg decitabine) Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) or the converse. In Courses ≥ 3, all participants received the FDC tablet Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
  Interventions: Drug: ASTX727 Fixed-Dose Combination

INTERVENTIONS:
Drug: ASTX727 Dose Escalation — Oral investigational product and approved IV decitabine
  Other Names: cedazuridine (E7727); oral decitabine; IV decitabine
  Arms: Phase 1 Dose Escalation
Drug: ASTX727 Dose Confirmation — Randomization cross over design for courses 1 and 2
  Other Names: ASTX727 oral (combination of oral E7727 and oral decitabine); IV decitabine
  Arms: Phase 2 Dose Confirmation
Drug: ASTX727 Fixed-Dose Combination — Fixed-dose investigational product
  Other Names: ASTX727 oral (combination of oral E7727 and oral decitabine)
  Arms: Phase 2 Fixed-Dose Combination

SUMMARY:
This first-in-human, 3-stage, open-label study evaluated the safety and pharmacokinetics of ASTX727, as well as determined the dose for later stages.

DETAILED DESCRIPTION:
The trial was designed to define daily doses of the individual components (cedazuridine [E7727] or decitabine) so that decitabine exposure after oral administration would be comparable to exposure after IV decitabine at the approved daily dose of 20 mg/m^2. The main objective of Phases 1 and 2 was to establish and confirm the doses of the 2 components to be used in the final fixed-dose combination (FDC) product (ASTX727) using mainly pharmacokinetics and pharmacodynamics as endpoints.

ELIGIBILITY:
Inclusion Criteria:

* International Prognostic Scoring System (IPSS) low, intermediate -1, intermediate-2, or high risk MDS (including chronic myelomonocytic leukemia; CMML) in Dose Escalation and Dose Confirmation-Randomization; only intermediate-2, or high risk MDS in Dose Confirmation-Open Label
* Eastern Cooperative Oncology Group (ECOG) 0 to 2
* No major surgery within 2 weeks of starting study treatment
* No cytotoxic chemotherapy within 2 weeks of starting study treatment
* Able to swallow pills

Exclusion Criteria:

* Previous treatment with 2 or more courses of decitabine (all stages) or azacitidine (Dose Confirmation stage only)
* Treatment with investigational therapy within 2 weeks of study treatment
* Uncontrolled medical disease(s) or active, uncontrolled infection
* Diagnosed with acute myeloid leukemia (AML)
* Active uncontrolled gastric or duodenal ulcer
* Known history of HIV or hepatitis C or B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Azab, MD, Study Director — Astex Pharmaceuticals, Inc.; James Lowder, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (17):
- United States (13):
  - Mayo Clinic, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Horizon Oncology, Lafayette, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center/ Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - M. D. Anderson, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Manero G, Griffiths EA, Steensma DP, Roboz GJ, Wells R, McCloskey J, Odenike O, DeZern AE, Yee K, Busque L, O'Connell C, Michaelis LC, Brandwein J, Kantarjian H, Oganesian A, Azab M, Savona MR. Oral cedazuridine/decitabine for MDS and CMML: a phase 2 pharmacokinetic/pharmacodynamic randomized crossover study. Blood. 2020 Aug 6;136(6):674-683. doi: 10.1182/blood.2019004143. PMID 32285126
- [Derived] Savona MR, Odenike O, Amrein PC, Steensma DP, DeZern AE, Michaelis LC, Faderl S, Harb W, Kantarjian H, Lowder J, Oganesian A, Azab M, Garcia-Manero G. An oral fixed-dose combination of decitabine and cedazuridine in myelodysplastic syndromes: a multicentre, open-label, dose-escalation, phase 1 study. Lancet Haematol. 2019 Apr;6(4):e194-e203. doi: 10.1016/S2352-3026(19)30030-4. PMID 30926081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase 1, 127 participants were screened and 44 were randomized and received at least one treatment. In Phase 2, a total of 138 were screened, 86 were randomized, and 80 received at least one treatment.
Pre-assignment Details: Response data for Phase 1 per June 2017 data cut and for Phase 2 per June 2018 data cut. Median follow up in Phase 1 was 1915.5 days (range: 1771-2213) and 1563.0 days in Phase 2 (range: 1199-1710).
Groups:
- Phase 1 Dose Escalation Cohort 1: Cohort 1 was administered 40 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 2: Cohort 2 was administered 60 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 3: Cohort 3 was administered 100 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 4: Cohort 4 was administered 100 mg oral cedazuridine and 40 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 5: Cohort 5 was administered 100 mg oral cedazuridine and 30 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 2 Dose Confirmation Sequence A: Participants were randomized in a 1:1 ratio to receive oral cedazuridine (100 mg) + decitabine (35 mg) capsules Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) in Sequence A. In Courses ≥ 3, all participants received cedazuridine and decitabine Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
- Phase 2 Dose Confirmation Sequence B: Participants were randomized in a 1:1 ratio to receive IV decibatine (20 mg/m^2) Dailyx5 in Course 1 followed by oral cedazuridine (100 mg) + decitabine (35 mg) capsules Dailyx5 in Course 2 (28 days per course) in Sequence B. In Courses ≥ 3, all participants received cedazuridine and decitabine Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
- Phase 2 Fixed-Dose Combination Sequence A: Participants were randomized in a 1:1 ratio to receive oral cedazuridine (100 mg) + decitabine (35 mg) tablets Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) in Sequence A. In Courses ≥ 3, all participants received cedazuridine and decitabine Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
- Phase 2 Fixed-Dose Combination Sequence B: Participants were randomized in a 1:1 ratio to receive IV decibatine (20 mg/m^2) Dailyx5 in Course 1 followed by oral cedazuridine (100 mg) + decitabine (35 mg) tablets Dailyx5 in Course 2 (28 days per course) in Sequence B. In Courses ≥ 3, all participants received cedazuridine and decitabine Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation Sequence A | Phase 2 Dose Confirmation Sequence B | Phase 2 Fixed-Dose Combination Sequence A | Phase 2 Fixed-Dose Combination Sequence B
Started | 7 | 6 | 6 | 6 | 19 | 25 | 25 | 16 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 6 | 6 | 19 | 25 | 25 | 16 | 14
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 1 | 1 | 5 | 15 | 14 | 10 | 11
Not completed — Progressive Disease | 2 | 1 | 2 | 0 | 9 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 3 | 2 | 0 | 3 | 8 | 8 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are shown for participants who received at least one dose of study drug.
Groups:
- Phase 2 Dose Confirmation: Participants were randomized in a 1:1 ratio to receive either oral cedazuridine (100 mg) + decitabine (35 mg) capsules Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) or the converse. In Courses ≥ 3, all participants received cedazuridine and decitabine capsules Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
- Phase 2 Fixed-Dose Combination: Participants were randomized in a 1:1 ratio to receive either the fixed-dose combination (FDC) tablet (100 mg cedazuridine/35 mg decitabine) Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2 (28 days per course) or the converse. In Courses ≥ 3, all participants received the FDC tablet Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19 | 50 | 30 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.1) | 72 (6.2) | 74 (4.8) | 75.2 (7.1) | 71.6 (8.8) | 69.7 (10.72) | 69.6 (10.57) | 70.6 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 2 | 4 | 9 | 10 | 33
  Male | 3 | 5 | 3 | 4 | 15 | 41 | 20 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 6
  Not Hispanic or Latino | 7 | 6 | 5 | 5 | 18 | 46 | 26 | 113
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 5
  White | 6 | 6 | 5 | 5 | 18 | 46 | 28 | 114
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 16
  United States | 7 | 6 | 6 | 6 | 19 | 42 | 22 | 108

OUTCOME MEASURES:

1. Primary Outcome: Mean Decitabine Area Under the Concentration Versus Time Curve (AUC0-t) on Day 5 by Cohort in Phase 1
Description: Mean AUC0-t of oral decitabine given with cedazuridine (E7727) following IV decitabine 20 mg/m^2 infusion on Day 5. AUCs were calculated by the linear up/log down method using the measured concentration-time values above the BQL (below the limit of quantification).
Time Frame: Day 5
Population: Participants who were successfully dosed according to criteria for both ASTX727 and IV decitabine dosing and with evaluable pharmacokinetic (PK) measurements are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 19
ng*h/mL | 53.6 (40) | 68.9 (44) | 94.8 (46) | 221 (74) | 146 (50)

2. Primary Outcome: Mean Decitabine Area Under the Plasma Concentration Versus Time Curve Ratio (5-day AUC0-t) in Phase 2
Description: Decitabine 5-day AUC ratio following IV decitabine 20 mg/m^2 infusion versus concomitant oral administration of decitabine + cedazuridine (E7727) or ASTX727 in the dose combination and fixed-dose combination stages, respectively. AUC0-t (the area under the concentration-time curve from time zero to the time of the last (tlast) quantifiable concentration (Ct)) by dose/cohort and course/days was used for estimating decitabine cumulative 5-day AUC0-t exposures.
Time Frame: Pre-dose to Day 5
Population: Participants with evaluable PK measurements are included. Phase 2 crossover design was used to compare AUC ratio for oral and IV administration.
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: Ratio of Geometric LSM
Groups:
- Phase 2 Dose Confirmation: Participants were randomized in a 1:1 ratio to receive either Sequence A: Oral cedazuridine (100 mg) + decitabine (35 mg) capsules Dailyx5 in Course 1 followed by IV decitabine (20 mg/m^2) Dailyx5 in Course 2; or Sequence B: IV decitabine (20 mg/m^2) Dailyx5 in Course 1 followed by cedazuridine + decitabine capsules Dailyx5 in Course 2 (28 days per course). In Courses ≥ 3, all participants received cedazuridine and decitabine capsules Dailyx5 in 28-day courses until disease progression, unacceptable toxicity, withdrawal of consent or withdrawal from the study.
Arm/Group | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 40 | 24
Ratio of Geometric LSM | 93.52 [82.10 to 106.50] | 97.59 [80.48 to 118.30]

3. Primary Outcome: Number of Participants With Dose-limiting Toxicity in Phase 1
Description: Number of participants with protocol-specified dose-limiting toxicities (DLTs) in the dose escalation stage. DLTs were defined using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAEv4.0), specifically ≥ Grade 3 non-hematologic toxicity (except Grade 3 nausea, vomiting, or diarrhea that is controllable by anti-emetics or optimal therapy or related to underlying disease or disease progression), specific Grade 3 laboratory tests, related prolonged Grade 4 thrombocytopenia or neutropenia that was not present prior to dosing, does not resolve within 14 days, and is not related to underlying disease, or any toxicity related to study treatment that results in treatment delays of >4 weeks after Day 28.
Time Frame: Up to Day 28 in Course 1 (28 days per course)
Population: The safety population includes participants in Phase 1 who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19
Participants | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Mean Maximum %LINE Demethylation in Phase 2
Description: Mean maximum % long interspread nuclear element-1 (LINE-1) demethylation after oral decitabine + cedazuridine (E7727) or ASTX727 (Course 1 or Course 2 - Treatment) compared with IV decitabine 20 mg/m^2 (Course 1 or Course 2 - IV Decitabine) in the dose confirmation and fixed-dose combination stages, respectively. Least squares mean of maximum %LINE-1 methylation change from baseline.
Time Frame: Pre-dose to Day 28 in Course 2 (28 days per course)
Population: The pharmacodynamic population includes all participants with evaluable data who received at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 48 | 30
Percent
  Course 1 - Treatment: number analyzed (Participants) | 24 | 16
  Course 1 - Treatment | 11.159 [9.023 to 13.294] | 10.077 [7.696 to 12.459]
  Course 1 - IV Decitabine: number analyzed (Participants) | 24 | 14
  Course 1 - IV Decitabine | 11.303 [9.167 to 13.439] | 12.665 [10.12 to 15.211]
  Course 2 - Treatment: number analyzed (Participants) | 22 | 9
  Course 2 - Treatment | 9.833 [7.446 to 12.219] | 8.134 [4.438 to 11.830]
  Course 2 - IV Decitabine: number analyzed (Participants) | 22 | 11
  Course 2 - IV Decitabine | 9.920 [7.534 to 12.307] | 8.230 [4.887 to 11.574]
Statistical Analysis 1: Comparison: Phase 2 Dose Confirmation; Test type: Equivalence — The 95% confidence intervals for the difference (oral - IV) were generated using an ANOVA model separately for Course 1 and Course 2; Mean Difference (Final Values) = -0.144, 95% CI 2-sided [-3.165 to 2.876] — Course 1
Statistical Analysis 2: Comparison: Phase 2 Dose Confirmation; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.087, 95% CI 2-sided [-3.463 to 3.288] — Course 2
Statistical Analysis 3: Comparison: Phase 2 Fixed-Dose Combination; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.588, 95% CI 2-sided [-6.074 to 0.899] — Course 1
Statistical Analysis 4: Comparison: Phase 2 Fixed-Dose Combination; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.096, 95% CI 2-sided [-5.080 to 4.888] — Course 2

5. Primary Outcome: Number of Participants With Overall Response in Phase 2
Description: The evaluation of response was based on International Working Group (IWG) 2006 MDS Response Criteria, with overall response calculated as number of participants with complete response+partial response+marrow complete response+hematological improvement (CR+PR+mCR+HI).
Time Frame: Up to approximately 29 months
Population: The efficacy population includes all participants in Phase 2 who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 50 | 30
Participants | 29 | 19

6. Secondary Outcome: Area Under the Concentration Versus Time Curve of Cedazuridine (E7727) and Cedazuridine-epimer
Description: AUC is a measure of the plasma concentration of the drug over time (AUC0-8). PK parameters are reported for the dose escalation stage by cohort in Phase 1 and dose confirmation and fixed-dose combination stages in Phase 2.
Time Frame: At specified timepoints from 0 to 24 hours post-dose
Population: Participants with evaluable PK measurements are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 37 | 19
ng*h/mL
  Cedazuridine: number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 32 | 14
  Cedazuridine | 1650 (43) | 1990 (64) | 3190 (53) | 4830 (51) | 3490 (46) | 2370 (56.8) | 1510 (49.4)
  Cedazuridine-epimer: number analyzed (Participants) | 6 | 6 | 5 | 3 | 12 | 37 | 19
  Cedazuridine-epimer | 503 (20) | 917 (64) | 1670 (48) | 2180 (34) | 1560 (56) | 1190 (48.3) | 710 (38)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cedazuridine (E7727) and Cedazuridine-epimer
Description: Cmax is the maximum observed plasma concentration. PK parameters are reported for the dose escalation stage by cohort in Phase 1 and dose confirmation and fixed-dose combination stages in Phase 2.
Time Frame: At specific timepoints from 0 to 24 hours post-dose
Population: Participants with evaluable PK measurements are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 47 | 29
ng/mL
  Cedazuridine | 309 (50) | 376 (67) | 636 (50) | 697 (75) | 570 (51) | 451 (51.4) | 293 (43.1)
  Cedazuridine-epimer | 96 (22) | 184 (70) | 343 (44) | 321 (47) | 291 (54) | 235 (49) | 154 (44.6)

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Cedazuridine (E7727) and Cedazuridine-epimer
Description: Tmax is the time to maximum observed plasma concentration. PK parameters are reported for the dose escalation stage by cohort in Phase 1 and the dose confirmation and fixed-dose combination stages in Phase 2.
Time Frame: At specific timepoints from 0 to 24 hours post-dose
Population: Participants with evaluable PK measurements are included.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 47 | 30
hours
  Cedazuridine: number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 47 | 29
  Cedazuridine | 3 [2 to 4] | 3 [2 to 4] | 3 [3 to 4] | 3 [2 to 6] | 3 [2 to 6] | 3 [1.50 to 4.08] | 3 [2.00 to 7.18]
  Cedazuridine-epimer: number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 47 | 29
  Cedazuridine-epimer | 3 [2 to 4] | 3 [2 to 3] | 3 [3 to 4] | 3 [2 to 6] | 3 [2 to 6] | 3 [1.50 to 6.17] | 3.05 [2.00 to 7.20]

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Decitabine
Description: Cmax is the maximum observed plasma concentration. PK parameters for plasma decitabine are reported for the dose escalation stage by cohort in Phase 1 and dose confirmation and fixed-dose combination stages in Phase 2.
Time Frame: At specific timepoints from 0 to 24 hours post-dose
Population: Participants with evaluable PK measurements are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 19 | 47 | 29
ng/mL | 54.0 (36) | 76.5 (42) | 80.9 (41) | 161 (51) | 138 (55) | 126 (70.9) | 126 (76.2)

10. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Decitabine in Phase 2
Description: Tmax is the time to reach maximum plasma concentration for decitabine. PK parameters for plasma decitabine are reported for the dose confirmation and fixed-dose combination stages.
Time Frame: At specific timepoints from 0 to 24 hours post-dose
Population: Participants with evaluable PK measurements are included.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 49 | 29
hours | 1.00 [0.47 to 3.00] | 0.95 [0.47 to 2.12]

11. Secondary Outcome: Duration of Complete Response in Phase 1
Description: Duration of response (in number of days) was calculated from the first time the response was observed to time of relapse or last time point in the study.
Time Frame: Up to 32 Months
Population: The efficacy population includes all participants in Phase 1 who received at least one dose of investigational product.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19
days | 546.00 [546.0 to 546.0] | 364.00 [56.0 to 672.0] | 470.00 [470.0 to 470.0] | 29.00 [29.0 to 29.0] | 399.0 [202.0 to 420.0]

12. Secondary Outcome: Duration of Complete Response in Phase 2 - Kaplan-Meier Estimate
Description: Duration of response (in number of days) was calculated from the first time the response was observed to time of relapse or last time point in the study. Kaplan-Meier estimate for complete response is shown.
Time Frame: Up to approximately 29 months
Population: The efficacy population includes all participants in Phase 2 who received at least one dose of investigational product.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 50 | 30
days | 413.0 [180.0 to 553.0] | 155.0 [35.0 to 285.0]

13. Secondary Outcome: Mean Maximum %LINE Demethylation in Phase 1
Description: Mean maximum % long interspread nuclear element-1 (LINE-1) demethylation decrease from baseline after oral decitabine + cedazuridine (E7727) or ASTX727 compared with IV decitabine 20 mg/m^2 in the dose escalation stage.
Time Frame: Pre-dose to Day 28 in Course 2 (28 days per course)
Population: The pharmacodynamic population includes all participants in Phase 1 with evaluable data who received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 18
Percent change
  Course 1 | -8.3 (5.28) | -9.2 (5.84) | -10.5 (7.55) | -12.1 (7.82) | -11.7 (5.67)
  Course 2 | -8.0 (3.56) | -7.1 (2.92) | -8.9 (5.42) | -8.6 (3.24) | -7.5 (5.47)

14. Secondary Outcome: Number of Participants With Overall Response in Phase 1
Description: The evaluation of response was based on International Working Group 2006 MDS Response Criteria, with overall response calculated as number of participants with complete response+partial response+marrow complete response+hematological improvement (CR+PR+mCR+HI).
Time Frame: Up to 32 months
Population: The efficacy population includes all participants in Phase 1 who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19
Participants | 4 | 3 | 2 | 1 | 3

15. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any treatment-emergent adverse event (AE) and any AE graded ≥3 using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 5 years
Population: The safety population includes all participants in Phase 1 and Phase 2 who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19 | 50 | 30
Participants
  Any Adverse Event | 6 | 6 | 6 | 6 | 19 | 50 | 30
  Any Grade ≥3 Adverse Event | 5 | 6 | 5 | 6 | 18 | 48 | 28

16. Secondary Outcome: Number of Participants With Hematological Improvement
Description: Hematological improvement was calculated as defined by the IWG 2006 MDS Response Criteria.
Time Frame: Up to 32 months
Population: The efficacy population includes all participants in Phase 1 and Phase 2 who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation Cohort 1: Cohort 1 was administered 40 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  ASTX727 Dose Escalation: Oral investigational product and approved IV decitabine
- Phase 1 Dose Escalation Cohort 2: Cohort 2 was administered 60 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  ASTX727 Dose Escalation: Oral investigational product and approved IV decitabine
- Phase 1 Dose Escalation Cohort 3: Cohort 3 was administered 100 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  ASTX727 Dose Escalation: Oral investigational product and approved IV decitabine
- Phase 1 Dose Escalation Cohort 4: Cohort 4 was administered 100 mg oral cedazuridine and 40 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  ASTX727 Dose Escalation: Oral investigational product and approved IV decitabine
- Phase 1 Dose Escalation Cohort 5: Cohort 5 was administered 100 mg oral cedazuridine and 30 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
  ASTX727 Dose Escalation: Oral investigational product and approved IV decitabine
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19 | 50 | 30
Participants | 4 | 3 | 2 | 0 | 3 | 8 | 7

17. Secondary Outcome: Number of Participants With Transfusion Independence
Description: Transfusion independence was calculated based on the number of transfusion-dependent participants at baseline who had no red blood cell or platelet transfusions for 56 consecutive days or more after treatment.
Time Frame: Up to 32 months
Population: The efficacy population includes all participants in Phase 1 and Phase 2 who received at least one dose of investigational product and were transfusion-dependent at baseline. Number analyzed is the number of participants who were transfusion-dependent at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation Cohort 5: Cohort 1 was administered 100 mg oral cedazuridine and 30 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 4 | 2 | 6 | 5 | 12 | 29 | 21
Participants
  Red Blood Cell: number analyzed (Participants) | 4 | 2 | 5 | 4 | 8 | 22 | 16
  Red Blood Cell | 2 | 0 | 3 | 0 | 2 | 11 | 8
  Platelet: number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 7 | 5
  Platelet | 0 | 0 | 1 | 0 | 1 | 3 | 3

18. Secondary Outcome: Number of Participants to Reach Acute Myeloid Leukemia (AML) or Death
Description: Number of participants to reach the event (AML or death), where time to reach AML was calculated as the number of days from the day the participant received the first dose of IV decitabine, oral decitabine + E7727, or the FDC tablet to the date of death or the date of MDS progression to AML as defined by ≥20% blasts in bone marrow or peripheral blood using the World Health Organization classification. Time to AML or death was censored on the last date of contact if a participant was lost to follow up prior to reaching a time-to-event endpoint.
Time Frame: Up to 32 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation Cohort 1: Starting cohort was administered 40 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 2: Starting cohort was administered 60 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 3: Starting cohort was administered 100 mg oral cedazuridine and 20 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 4: Starting cohort was administered 100 mg oral cedazuridine and 40 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
- Phase 1 Dose Escalation Cohort 5: Starting cohort was administered 100 mg oral cedazuridine and 30 mg oral decitabine. Participants were enrolled into successive cohorts in which either the cedazuridine or decitabine oral dose was varied in Course 1 Day 2 through Course 1 Day 5 for comparison with a single dose of IV decitabine at 20 mg/m^2 administered on Day 1 by continuous IV infusion over 1 hour (28 days per course).
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19 | 50 | 30
Participants
  Censored | 4 | 5 | 6 | 5 | 11 | 22 | 11
  Event | 3 | 1 | 0 | 1 | 8 | 28 | 19

19. Secondary Outcome: Number of Participants With Overall Survival
Description: Overall survival was defined as the number of days from the day the participant received the first dose of IV decitabine, oral decitabine + E7727, or the FDC tablet to the date of death, regardless of cause.
Time Frame: Up to 32 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 19 | 50 | 30
Participants
  Censored | 6 | 5 | 6 | 5 | 15 | 26 | 14
  Event | 1 | 1 | 0 | 1 | 4 | 24 | 16

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Treatment-emergent adverse events were recorded from the start of study treatment until 30 days after the last dose of study treatment.
Arm/Group | Phase 1 Dose Escalation Cohort 1 | Phase 1 Dose Escalation Cohort 2 | Phase 1 Dose Escalation Cohort 3 | Phase 1 Dose Escalation Cohort 4 | Phase 1 Dose Escalation Cohort 5 | Phase 2 Dose Confirmation | Phase 2 Fixed-Dose Combination
All-Cause Mortality (participants affected / at risk) | 2/7 | 2/6 | 1/6 | 1/6 | 5/19 | 29/50 | 21/30
Serious Adverse Events (participants affected / at risk) | 2/7 | 4/6 | 2/6 | 6/6 | 14/19 | 39/50 | 25/30
Other Adverse Events (participants affected / at risk) | 6/7 | 6/6 | 6/6 | 6/6 | 18/19 | 48/50 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation Cohort 1 (N=7) | Phase 1 Dose Escalation Cohort 2 (N=6) | Phase 1 Dose Escalation Cohort 3 (N=6) | Phase 1 Dose Escalation Cohort 4 (N=6) | Phase 1 Dose Escalation Cohort 5 (N=19) | Phase 2 Dose Confirmation (N=50) | Phase 2 Fixed-Dose Combination (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (5) | 1 (1) | 1 (1) | 2 (8) | 2 (2) | 17 (31) | 7 (10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (3) | 8 (8) | 5 (6)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 8 (8)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mental status change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alpha hemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation Cohort 1 (N=7) | Phase 1 Dose Escalation Cohort 2 (N=6) | Phase 1 Dose Escalation Cohort 3 (N=6) | Phase 1 Dose Escalation Cohort 4 (N=6) | Phase 1 Dose Escalation Cohort 5 (N=19) | Phase 2 Dose Confirmation (N=50) | Phase 2 Fixed-Dose Combination (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (16) | 3 (4) | 4 (11) | 3 (7) | 10 (34) | 27 (67) | 15 (59)
Neutropenia (Blood and lymphatic system disorders) | 3 (13) | 2 (12) | 4 (4) | 1 (4) | 6 (24) | 28 (125) | 12 (53)
Anemia (Blood and lymphatic system disorders) | 4 (8) | 1 (1) | 2 (2) | 3 (6) | 5 (16) | 16 (46) | 8 (23)
Leukopenia (Blood and lymphatic system disorders) | 1 (6) | 2 (6) | 1 (2) | 0 (0) | 4 (24) | 12 (47) | 11 (45)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 5 (6)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 2 (4) | 7 (8) | 17 (24) | 12 (15)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (4) | 3 (3) | 3 (4) | 5 (6) | 13 (20) | 14 (18)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (2) | 2 (3) | 1 (2) | 1 (1) | 19 (28) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 4 (5) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 6 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 3 (3) | 8 (10)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (4) | 5 (7) | 3 (4) | 5 (7) | 6 (6) | 23 (37) | 12 (15)
Edema peripheral (General disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 4 (4) | 13 (16) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 7 (13) | 7 (9)
Edema (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 7 (8) | 9 (12)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 3 (4)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heliobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 6 (7) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (8) | 4 (5)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (2) | 1 (1) | 1 (1) | 5 (10) | 11 (22) | 4 (9)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 7 (10) | 6 (7)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 8 (10) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 2 (3) | 0 (0) | 2 (4) | 4 (8) | 9 (18) | 3 (5)
Blood bilirubin increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 5 (9) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 6 (11) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Electrocardiogram repolarization abnormality (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (5) | 3 (4) | 2 (3) | 12 (23) | 5 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 5 (9) | 10 (13) | 6 (12)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (5) | 5 (6) | 6 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 5 (5) | 7 (16) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 6 (13) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 3 (3) | 8 (12) | 7 (8)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 4 (7) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 10 (13) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (5) | 11 (15) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 12 (15) | 10 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 4 (6)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (4) | 6 (12) | 7 (7)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 14 (19) | 13 (14)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoasthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 6 (7) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 12 (14) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 12 (15) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 6 (7) | 6 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (15) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 4 (5) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 5 (5)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gasdtroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02103478/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02103478/SAP_001.pdf